CLINICAL TRIAL: NCT03765606
Title: The Bioavailability of Cocoa Flavan-3-ols and Interaction With the Methylxanthine, Theobromine: a Study With Ileostomists
Brief Title: Cocoa Ileostomy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UREC/18/0007
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-06

CONDITIONS: Ileostomy - Stoma
Keywords: Cocoa Flavan-3-ols; methylaxanthin; theobromine; Ileostomists; bioavailability; randomised controlled trial

STUDY DESIGN:
Intervention Model Description: Randomised double-blinded crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cocoa Flavanol beverage mix (Placebo Comparator): Cocoa Flavanol beverage mix (flavanols, 566mg; caffeine, 11mg & theobromine, 93mg)
  Interventions: Dietary Supplement: Cocoa Flavanol beverage mix
- De-xanthinated Cocoa Flavanol beverage mix (Experimental): De-xanthinated Cocoa Flavanol beverage mix (flavanols, 583mg; caffeine, 0.6mg & theobromine, 0.2mg)
  Interventions: Dietary Supplement: De-xanthinated Cocoa Flavanol beverage mix

INTERVENTIONS:
Dietary Supplement: Cocoa Flavanol beverage mix — Acute consumption of single portion of cocoa powder dissolved in 310g 1% milk.
  Arms: Cocoa Flavanol beverage mix
Dietary Supplement: De-xanthinated Cocoa Flavanol beverage mix — Acute consumption of single portion of cocoa powder dissolved in 310g 1% milk.
  Arms: De-xanthinated Cocoa Flavanol beverage mix

SUMMARY:
There is substantial interest in the potential role of chocolate and its primary bioactive component; flavan-3-ol, (-)-epicatechin, in both the prevention and management of cardiovascular disease (CVD). Numerous observational studies have found the association between high cocoa intake and a reduced CVD risk and mortality, yet the impact of these mechanisms in vivo is unclear. In order to have a beneficial effect, these cocoa flavan-3-ols must be absorbed in the body in a forms, while still maintaining its advantageous characteristics. Consumption studies with ileostomists who have had their colon removed,provide information regarding the bioavailability and bioactivity of (-)-epicatechin and flavan-3-ols from cocoa, therefore the aim of this study is to determine the impact of methylaxanthines (including theobromine) on bioavailability of cocoa flavan-3-ols prior to entering the colon.

This study has a randomised double blinded crossover control design, being applied to ileostomy patients who are aged 18-65 years, N=10, 5 per group. The study is divided into two phases. During the first phase, subjects will partake in a 2-day restriction diet (No phenolic foods) and an overnight fast prior to sampling. Ileal fluid (0hr) is obtained from participants. They will then be asked to consume the cocoa flavanol beverage dissolved in 310g 1% milk. After this urine and ieal fluid is collected every 4 hours at 3 more time points and blood every hour at 8 time points. A 24 hr urine and ieal fluid sample is collected the following day. There will be a 1-week wash out period between each phase. Procedure is repeated again for phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Undergone an ileostomy and be more than 1.5-years post-operative
* Male or female
* Aged between 18-65 years
* Non-smoking
* Not lactose/milk/dairy intolerant

Exclusion Criteria:

* Has not undergone an ileostomy and/or is less than 1.5 year post-operative
* Pregnant/ lactating females
* Smokers
* Lactose/milk/diary intolerant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
cocoa flavan-3-ols bio-availability | 24-hour period post-consumption
  Recovery of ingested flavan-3-ols in ileal fluid
cocoa flavan-3-ols bio-availability | Change over 8-hour period post-consumption
  Uptake of ingested flavan-3-ols in plasma
cocoa flavan-3-ols availability | Change over 24-hour period post-consumption
  Recovery of ingested flavan-3-ols in urine

SECONDARY OUTCOMES:
Simulated gut microbiota | Change over 24-hour in vitro fermentation period
  Ileal fluid with/without simulated colonic fermentation

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ottaviani JI, Fong RY, Borges G, Kimball J, Ensunsa JL, Medici V, Pourshahidi LK, Kane E, Ward K, Durkan R, Dobani S, Lawther R, O'Connor G, Gill CIR, Schroeter H, Crozier A. Flavan-3-ol-methylxanthine interactions: Modulation of flavan-3-ol bioavailability in volunteers with a functional colon and an ileostomy. Free Radic Biol Med. 2023 Feb 20;196:1-8. doi: 10.1016/j.freeradbiomed.2023.01.003. Epub 2023 Jan 5. PMID 36621554